CLINICAL TRIAL: NCT00373256
Title: A Phase 3 Study Of SU011248 In Combination With Paclitaxel Versus Bevacizumab With Paclitaxel In The First-Line Advanced Disease Setting In Patients Having Breast Cancer
Brief Title: A Study Of SU011248 Plus Paclitaxel Versus Bevacizumab Plus Paclitaxel In Patients With Advanced Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6181094
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2010-10-08 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Breast Neoplasms
Keywords: Breast cancer; advanced; sunitinib; bevacizumab; paclitaxel; Phase 3
MeSH Terms: conditions — Breast Neoplasms | interventions — Sunitinib; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Sunitinib; Drug: paclitaxel
- B (Active Comparator)
  Interventions: Drug: bevacizumab; Drug: paclitaxel

INTERVENTIONS:
Drug: Sunitinib — Sunitinib 25 mg daily by oral capsules with titration up to 37.5 mg,
  Other Names: SU011248, Sutent
  Arms: A
Drug: paclitaxel — Paclitaxel 90 mg/m2 IV, 3 weekly doses every 28 days until progression or unacceptable toxicity.
  Arms: A
Drug: bevacizumab — Bevacizumab 10 mg/kg IV every 2 weeks.
  Other Names: Avastin
  Arms: B
Drug: paclitaxel — Paclitaxel 90 mg/m2 IV, 3 weekly doses every 28 days until progression or unacceptable toxicity.
  Arms: B

SUMMARY:
To compare treatment with SU011248 plus paclitaxel versus bevacizumab plus paclitaxel to determine which treatment works better against breast cancer

DETAILED DESCRIPTION:
On May 27, 2009, the independent Data Monitoring Committee (DMC) reviewed the progress of Study A6181094. The DMC determined Study A6181094 had met pre-specified futility criteria and was unlikely to meet its primary endpoint to demonstrate a statistically significant improvement in progression-free survival (PFS) in patients treated with sunitinib plus paclitaxel versus bevacizumab plus paclitaxel. Pfizer notified clinical trial investigators involved in the study and regulatory agencies of these findings. Enrollment in this study has been stopped.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced breast cancer.
* Measurable disease as per RECIST (Response Evaluation Criterion) in Solid Tumors or bone-only disease.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1.

Exclusion Criteria:

* No prior treatment with cytotoxics in the advanced disease setting.
* HER2/neu positive disease unless trastuzumab was previously received or is contraindicated.
* Treatment with a taxane in the adjuvant setting unless disease free interval >12 months after end of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (193):
- United States (184):
  - Pfizer Investigational Site, Bessemer, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Daphne, Alabama
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Flagstaff, Arizona
  - Pfizer Investigational Site, Sedona, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Antioch, California
  - Pfizer Investigational Site, Baldwin Park, California
  - Pfizer Investigational Site, Bellflower, California
  - Pfizer Investigational Site, Fontana, California
  - Pfizer Investigational Site, Fountain Valley, California
  - Pfizer Investigational Site, Gilroy, California
  - Pfizer Investigational Site, Hawthorne, California
  - Pfizer Investigational Site, Hayward, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Long Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Martinez, California
  - Pfizer Investigational Site, Milpitas, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, Mountain View, California
  - Pfizer Investigational Site, Oakland, California
  - Pfizer Investigational Site, Ontario, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Oxnard, California
  - Pfizer Investigational Site, Panorama City, California
  - Pfizer Investigational Site, Pinole, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, San Jose, California
  - Pfizer Investigational Site, San Sacramento, California
  - Pfizer Investigational Site, Santa Clara, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Union City, California
  - Pfizer Investigational Site, Vallejo, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Woodland Hills, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Lakewood, Colorado
  - Pfizer Investigational Site, Littleton, Colorado
  - Pfizer Investigational Site, Lone Tree, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Parker, Colorado
  - Pfizer Investigational Site, Thornton, Colorado
  - Pfizer Investigational Site, Norwalk, Connecticut
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Coral Springs, Florida
  - Pfizer Investigational Site, Davie, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Inverness, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Columbus, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Macon, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Harvey, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Tinley Park, Illinois
  - Pfizer Investigational Site, Vernon Hills, Illinois
  - Pfizer Investigational Site, Avon, Indiana
  - Pfizer Investigational Site, Beech Grove, Indiana
  - Pfizer Investigational Site, Carmel, Indiana
  - Pfizer Investigational Site, Fishers, Indiana
  - Pfizer Investigational Site, Greenfield, Indiana
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Mooresville, Indiana
  - Pfizer Investigational Site, Munster, Indiana
  - Pfizer Investigational Site, New Albany, Indiana
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Annapolis, Maryland
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Randallstown, Maryland
  - Pfizer Investigational Site, Burlington, Massachusetts
  - Pfizer Investigational Site, Peabody, Massachusetts
  - Pfizer Investigational Site, Coon Rapids, Minnesota
  - Pfizer Investigational Site, Robbinsdale, Minnesota
  - Pfizer Investigational Site, Ocean Springs, Mississippi
  - Pfizer Investigational Site, Pascagoula, Mississippi
  - Pfizer Investigational Site, Columbia, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Lee's Summit, Missouri
  - Pfizer Investigational Site, Fremont, Nebraska
  - Pfizer Investigational Site, Grand Island, Nebraska
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Corning, New York
  - Pfizer Investigational Site, Jamaica, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Clinton, North Carolina
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Goldsboro, North Carolina
  - Pfizer Investigational Site, Hickory, North Carolina
  - Pfizer Investigational Site, Kenansville, North Carolina
  - Pfizer Investigational Site, Kinston, North Carolina
  - Pfizer Investigational Site, Lenoir, North Carolina
  - Pfizer Investigational Site, Pollocksville, North Carolina
  - Pfizer Investigational Site, Raleight, North Carolina
  - Pfizer Investigational Site, Raliegh, North Carolina
  - Pfizer Investigational Site, Richlands, North Carolina
  - Pfizer Investigational Site, Washington, North Carolina
  - Pfizer Investigational Site, Wilson, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Canton, Ohio
  - Pfizer Investigational Site, Dover, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Springfield, Oregon
  - Pfizer Investigational Site, Tualatin, Oregon
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Ephrata, Pennsylvania
  - Pfizer Investigational Site, Hershey, Pennsylvania
  - Pfizer Investigational Site, Kingston, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Sayre, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Easley, South Carolina
  - Pfizer Investigational Site, Greenville, South Carolina
  - Pfizer Investigational Site, Seneca, South Carolina
  - Pfizer Investigational Site, Spartanburg, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Amarillo, Texas
  - Pfizer Investigational Site, Antonio, Texas
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Bedford, Texas
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Forth Worth, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Kerrville, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, Midland, Texas
  - Pfizer Investigational Site, Round Rock, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, San Marcos, Texas
  - Pfizer Investigational Site, Shenandoah, Texas
  - Pfizer Investigational Site, Tyler, Texas
  - Pfizer Investigational Site, Waco, Texas
  - Pfizer Investigational Site, Ogden, Utah
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Christiansburg, Virginia
  - Pfizer Investigational Site, Fairfax, Virginia
  - Pfizer Investigational Site, Leesburg, Virginia
  - Pfizer Investigational Site, Norton, Virginia
  - Pfizer Investigational Site, Roanoke, Virginia
  - Pfizer Investigational Site, Salem, Virginia
  - Pfizer Investigational Site, Woodbridge, Virginia
  - Pfizer Investigational Site, Wytheville, Virginia
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Kennewick, Washington
  - Pfizer Investigational Site, Lakewood, Washington
  - Pfizer Investigational Site, Moses Lake, Washington
  - Pfizer Investigational Site, Puyallup, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Vancouver, Washington
  - Pfizer Investigational Site, Wenatchee, Washington
  - Pfizer Investigational Site, Huntington, West Virginia
  - Pfizer Investigational Site, Morgantown, West Virginia
- Germany (3):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Trier
- Italy (3):
  - Pfizer Investigational Site, Cremona
  - Pfizer Investigational Site, Grosseto
  - Pfizer Investigational Site, Olbia
- Spain (3):
  - Pfizer Investigational Site, Cabueñes, Gijon
  - Pfizer Investigational Site, Guadalajara, Guadalajara
  - Pfizer Investigational Site, Madrid, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181094&StudyName=A%20Study%20Of%20SU011248%20Plus%20Paclitaxel%20Versus%20Bevacizumab%20Plus%20Paclitaxel%20In%20Patients%20With%20Advanced%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib + Paclitaxel: Starting sunitinib doses of 25 milligrams (mg) daily. After Cycle 1, escalation to 37.5 mg daily was permitted in the absence of complicated neutropenia and if all 3 Cycle 1 paclitaxel doses were successfully administered at 90 milligrams per square meter (mg/m^2), at discretion of the investigator. Paclitaxel could have been reduced to 65 mg/m^2 based on tolerability; re-escalation to 80 or 90 mg/m^2 upon recovery was permitted.
- Bevacizumab + Paclitaxel: Bevacizumab 10 milligrams per kilogram (mg/kg); infusion duration according to standard of care. Paclitaxel starting dose of 90 mg/m^2, as a 1 hour infusion. Paclitaxel could have been reduced to 65 mg/m^2 based on tolerability; re-escalation to 80 or 90 mg/m^2 upon recovery was permitted.
Period: Overall Study
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Started | 241 | 247
Treated | 235 | 236
Completed | 0 | 0
Not Completed | 241 | 247
Not completed — Adverse Event (AE) | 1 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 9 | 8
Not completed — Objective Progression or Relapse | 111 | 104
Not completed — Refused Treatment-Reason Other Than AE | 4 | 7
Not completed — Other | 73 | 107
Not completed — Protocol Violation | 0 | 2
Not completed — Study Terminated by Sponsor | 41 | 13

BASELINE CHARACTERISTICS:
Groups:
- Sunitinib + Paclitaxel: Starting sunitinib doses of 25 mg daily. After Cycle 1, escalation to 37.5 mg daily was permitted in the absence of complicated neutropenia and if all 3 Cycle 1 paclitaxel doses were successfully administered at 90 mg/m^2, at discretion of the investigator. Paclitaxel could have been reduced to 65 mg/m^2 based on tolerability; re-escalation to 80 or 90 mg/m^2 upon recovery was permitted.
- Bevacizumab + Paclitaxel: Bevacizumab 10 mg/kg; infusion duration according to standard of care. Paclitaxel starting dose of 90 mg/m^2, as a 1 hour infusion. Paclitaxel could have been reduced to 65 mg/m^2 based on tolerability; re-escalation to 80 or 90 mg/m^2 upon recovery was permitted.
- Total: Total of all reporting groups
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel | Total
Number analyzed (Participants) | 241 | 247 | 488
Age, Customized [Number; unit: Participants]
  18 to 44 years | 38 | 40 | 78
  45 to 64 years | 144 | 137 | 281
  more than 65 years | 59 | 70 | 129
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 247 | 487
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Time from date of randomization to the date of the first documentation of objective tumor progression or death due to any cause, whichever occurred first. PFS = (first event date minus randomization date +1) divided by 30.4
Time Frame: From date of randomization through Day 1 and every 8 weeks thereafter up to 18 months or death
Population: The intent-to-treat (ITT) population included all patients who were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 242 | 243
Months | 7.4 [6.9 to 8.5] | 9.2 [7.7 to 13.0]
Statistical Analysis 1: Comparison: Sunitinib + Paclitaxel vs Bevacizumab + Paclitaxel; Test type: Superiority or Other; p = 0.9986, Log Rank — p-value from 1-sided log-rank stratified for prior adjuvant chemotherapy, hormone receptor status, disease-free interval from prior adjuvant treatment. Stratification factors from Interactive Voice Randomization System; Hazard Ratio (HR) = 1.6299, 95% CI 2-sided [1.1793 to 2.2527] — Assuming proportional hazards, a hazard ratio greater than 1 indicated a reduction in hazard rate in favor Bevacizumab + Paclitaxel

2. Secondary Outcome: Number of Participants With Objective Response
Description: Objective response = participants with confirmed complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST). A CR was defined as the disappearance of all target lesions. A PR was defined as a > = 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From date of randomization through Day 1 and every 8 weeks thereafter up to 18 months
Population: ITT
Measure: Number; unit: participants
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 242 | 243
participants | 78 | 78
Statistical Analysis 1: Comparison: Sunitinib + Paclitaxel; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 32.2, 95% CI 2-sided [26.4 to 38.5]
Statistical Analysis 2: Comparison: Bevacizumab + Paclitaxel; Test type: Superiority or Other; Objective Response Rate (ORR) (percent) = 32.1, 95% CI 2-sided [26.3 to 38.4]

3. Secondary Outcome: Duration of Response (DR)
Description: DR=time from the first documentation of objective tumor response (CR or PR) that was subsequently confirmed to first documentation of objective disease progression or death due to any cause, whichever was first. DR was calculated as [the date response ended (ie, date of progressive disease or death) minus first CR or PR date that was subsequently confirmed +1)] divided by 30.4.
Time Frame: From date of randomization through Day 1 and every 8 weeks thereafter up to 18 months or death due to any cause
Population: ITT. DR was calculated for the subgroup of subjects with objective response. 78 subjects reported CR or PR response and were analyzed for DR in each treatment group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 78 | 78
Months | 6.3 [5.6 to 7.9] | 14.8 [7.4 to 21.7]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from date of randomization to death due to any cause. OS (in months) was calculated as (date of death minus randomization date +1) divided by 30.4.
Time Frame: From date of randomization up to 5 years. Survival follow-up changed to 28-days after treatment discontinuation when study was discontinued.
Population: ITT. The median OS for bevacizumab + paclitaxel at the time of data cut off was not reached; therefore, it could not be calculated.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 242 | 243
Months | 17.6 [16.4 to NA] — The upper confidence interval was not reached. | NA [22.1 to NA] — The median OS for bevacizumab + paclitaxel at the time of data cut off was not reached; therefore, it could not be calculated.

5. Secondary Outcome: Percentage of Participants Surviving at 1 and 2 Years
Description: Percentage of those surviving at the end of one year or end of 2 years from the first dose of study treatment.
Time Frame: Year 1, Year 2
Population: ITT.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 242 | 243
percentage of participants
  Year 1 | 76.8 | 83.7
  Year 2 | 35.5 | 61.0
Statistical Analysis 1: Comparison: Sunitinib + Paclitaxel; 1 year; Test type: Superiority or Other; Percentage = 76.8, 95% CI 2-sided [68.7 to 83.0]
Statistical Analysis 2: Comparison: Sunitinib + Paclitaxel; 2 years; Test type: Superiority or Other; Percentage = 35.5, 95% CI 2-sided [20.9 to 50.3]
Statistical Analysis 3: Comparison: Bevacizumab + Paclitaxel; 1 year; Test type: Superiority or Other; Percentage = 83.7, 95% CI 2-sided [76.0 to 89.1]
Statistical Analysis 4: Comparison: Bevacizumab + Paclitaxel; 2 years; Test type: Superiority or Other; Percentage = 61.0, 95% CI 2-sided [43.2 to 74.7]

6. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30)
Description: EORTC QLQ-C30: global health/QoL, functional domains (physical, role, cognitive, emotional, social), and symptom scales/items (fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea). Recall period: past week; response range: not at all to very much, global/QOL range: very poor to excellent. Scale score range: 0 to 100. Higher functional/global QoL score = better functioning and higher symptom score = greater degree of symptoms.
Time Frame: Day 1 of Cycles 1 through 7 and then odd-numbered cycles thereafter until 18 months
Population: ITT. EORTC QLQ-C30 evaluations were not analyzed since enrollment in this study was terminated early for futility.
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: EORTC QLQ Breast Cancer Module (BR23)
Description: BR23: measured disease related symptoms of dry mouth, eye pain, hair loss, hot flushes, attractiveness, future health, sexual activity, arm/shoulder pain, breast pain, swollen breast, and skin problems on the breast. Recall period: past week; response range: not at all to very much. Scale score range: 0 to 100. Higher symptom score = greater degree of symptoms.
Time Frame: Day 1 of Cycles 1 through 7 and then odd-numbered cycles thereafter until 18 months
Population: ITT. BR23 evaluations were not analyzed since enrollment in this study was terminated early for futility at the first interim analysis.
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Euro Quality of Life-5 Dimension (EQ-5D)
Description: EQ-5D: health status in 5 dimensions (mobility, self-care, pain/discomfort, anxiety/depression, usual activities). Three-level scale (1=no problem, 2=some problem, and 3=extreme problem). A single score between 1 and 3 is generated for each domain. For each subject, the outcome rating on the 5 domains could be mapped to a single index through an algorithm. The index ranges between 0 and 1, with the higher score indicating a better health state perceived by the subject.
Time Frame: Day 1 of Cycles 1 through 7 and then odd-numbered cycles thereafter until 18 months
Population: ITT. EQ-5D evaluations were not analyzed since enrollment in this study was terminated early for futility at the first interim analysis.
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: EQ - Visual Analog Scale (EQ-VAS)
Description: EQ-VAS score on the self-rated "thermometer," indicating the patient's own assessment of their health status from 0 (worst) to 100 (best) imaginable health state.
Time Frame: Day 1 of Cycles 1 through 7 and then odd-numbered cycles thereafter until 18 months
Population: ITT. EQ-VAS evaluations were not analyzed since enrollment in this study was terminated early for futility at the first interim analysis.
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Biomarkers
Description: Concentrations of plasma proteins (eg, soluble Vascular Endothelial Growth Factor Receptor 2 [VEGFR2] and VEGFR3, VEGF-A, placental growth factor [PlGF], soluble KIT, and possibly soluble PDGFRβ and PDGF) that may be associated with angiogenesis and tumor proliferation.
Time Frame: Day 1 of Cycles 1 through 3 and 5, Day 8 of Cycle 1, and Day 15 of Cycle 1
Population: ITT. Biomarker data were collected, but since the study was stopped early and there were too few events of OS, PFS, etc, data were not analyzed.
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib + Paclitaxel | Bevacizumab + Paclitaxel
Serious Adverse Events (participants affected / at risk) | 89/235 | 85/242
Other Adverse Events (participants affected / at risk) | 232/235 | 239/242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sunitinib + Paclitaxel (N=235) | Bevacizumab + Paclitaxel (N=242)
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 0
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 1
Asthenia (General disorders) | 3 | 2
Chest pain (General disorders) | 2 | 0
Disease progression (General disorders) | 7 | 7
Fatigue (General disorders) | 2 | 2
General physical health deterioration (General disorders) | 4 | 2
Generalised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 4 | 5
Cholecystitis (Hepatobiliary disorders) | 3 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 3 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 2
Neutropenic sepsis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 3 | 4
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 3
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 2
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 3 | 5
Viral diarrhoea (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Ammonia increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0/236
Dehydration (Metabolism and nutrition disorders) | 15 | 12
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 2
Myelitis transverse (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 5
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mastectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0
Arterial rupture (Vascular disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib + Paclitaxel (N=235) | Bevacizumab + Paclitaxel (N=242)
Anaemia (Blood and lymphatic system disorders) | 104 | 65
Leukopenia (Blood and lymphatic system disorders) | 63 | 55
Lymphopenia (Blood and lymphatic system disorders) | 17 | 13
Neutropenia (Blood and lymphatic system disorders) | 170 | 98
Thrombocytopenia (Blood and lymphatic system disorders) | 56 | 15
Lacrimation increased (Eye disorders) | 14 | 14
Vision blurred (Eye disorders) | 15 | 9
Abdominal pain (Gastrointestinal disorders) | 34 | 36
Abdominal pain upper (Gastrointestinal disorders) | 21 | 7
Constipation (Gastrointestinal disorders) | 69 | 92
Diarrhoea (Gastrointestinal disorders) | 145 | 109
Dry mouth (Gastrointestinal disorders) | 15 | 12
Dyspepsia (Gastrointestinal disorders) | 41 | 31
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 28 | 12
Haemorrhoids (Gastrointestinal disorders) | 14 | 10
Nausea (Gastrointestinal disorders) | 118 | 113
Oral pain (Gastrointestinal disorders) | 21 | 8
Stomatitis (Gastrointestinal disorders) | 44 | 23
Vomiting (Gastrointestinal disorders) | 67 | 58
Asthenia (General disorders) | 29 | 21
Chest pain (General disorders) | 12 | 10
Chills (General disorders) | 13 | 17
Fatigue (General disorders) | 148 | 156
Mucosal inflammation (General disorders) | 50 | 52
Oedema (General disorders) | 11 | 11
Oedema peripheral (General disorders) | 39 | 33
Pain (General disorders) | 25 | 17
Pyrexia (General disorders) | 43 | 40
Sinusitis (Infections and infestations) | 18 | 21
Upper respiratory tract infection (Infections and infestations) | 20 | 45
Urinary tract infection (Infections and infestations) | 31 | 43
Alanine aminotransferase increased (Investigations) | 29 | 12
Aspartate aminotransferase increased (Investigations) | 26 | 16
Blood alkaline phosphatase increased (Investigations) | 21 | 11
Weight decreased (Investigations) | 32 | 30
Decreased appetite (Metabolism and nutrition disorders) | 71 | 62
Dehydration (Metabolism and nutrition disorders) | 31 | 22
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 30
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 39 | 27
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 19
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 64
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 39
Bone pain (Musculoskeletal and connective tissue disorders) | 30 | 26
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 15
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9 | 17
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 | 21
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 42
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 54
Dizziness (Nervous system disorders) | 24 | 51
Dysgeusia (Nervous system disorders) | 62 | 53
Headache (Nervous system disorders) | 56 | 67
Neuropathy peripheral (Nervous system disorders) | 93 | 116
Paraesthesia (Nervous system disorders) | 16 | 18
Peripheral sensory neuropathy (Nervous system disorders) | 21 | 32
Anxiety (Psychiatric disorders) | 31 | 23
Depression (Psychiatric disorders) | 19 | 23
Insomnia (Psychiatric disorders) | 50 | 48
Cough (Respiratory, thoracic and mediastinal disorders) | 46 | 72
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 | 63
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 69 | 100
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 18
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 32
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 116 | 142
Dry skin (Skin and subcutaneous tissue disorders) | 25 | 9
Erythema (Skin and subcutaneous tissue disorders) | 14 | 10
Nail disorder (Skin and subcutaneous tissue disorders) | 12 | 50
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 29 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 18 | 21
Rash (Skin and subcutaneous tissue disorders) | 66 | 60
Flushing (Vascular disorders) | 15 | 12
Hot flush (Vascular disorders) | 20 | 20
Hypertension (Vascular disorders) | 52 | 77
Hypotension (Vascular disorders) | 15 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 4
Granulocytopenia (Blood and lymphatic system disorders) | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Macrocytosis (Blood and lymphatic system disorders) | 2 | 0
Microcytosis (Blood and lymphatic system disorders) | 0 | 1
Neutrophilia (Blood and lymphatic system disorders) | 2 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 4
Cardiomegaly (Cardiac disorders) | 0 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 1
Cyanosis (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 4 | 5
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 6
Pericardial effusion (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 2
Splinter haemorrhages (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 8 | 12
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 2 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 5 | 3
Tinnitus (Ear and labyrinth disorders) | 3 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 4
Cushingoid (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 6 | 7
Blindness unilateral (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 3 | 0
Conjunctival oedema (Eye disorders) | 1 | 0
Conjunctival pallor (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 5 | 7
Dacryostenosis acquired (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 5 | 2
Dry eye (Eye disorders) | 4 | 6
Eye disorder (Eye disorders) | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 0
Eye irritation (Eye disorders) | 2 | 1
Eye pain (Eye disorders) | 1 | 2
Eye pruritus (Eye disorders) | 0 | 2
Eye swelling (Eye disorders) | 1 | 0
Eyelid oedema (Eye disorders) | 4 | 0
Eyelid ptosis (Eye disorders) | 1 | 0
Eyelids pruritus (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Halo vision (Eye disorders) | 1 | 0
Keratoconjunctivitis sicca (Eye disorders) | 0 | 1
Mydriasis (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Periorbital oedema (Eye disorders) | 2 | 1
Photophobia (Eye disorders) | 0 | 1
Pupils unequal (Eye disorders) | 1 | 1
Retinopathy hypertensive (Eye disorders) | 0 | 1
Scotoma (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 4
Visual impairment (Eye disorders) | 1 | 6
Vitreous floaters (Eye disorders) | 2 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 4 | 8
Abdominal pain lower (Gastrointestinal disorders) | 4 | 3
Abdominal tenderness (Gastrointestinal disorders) | 4 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 2
Anorectal discomfort (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 3 | 5
Chapped lips (Gastrointestinal disorders) | 2 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 1
Cheilosis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 | 0
Diverticulum (Gastrointestinal disorders) | 2 | 1
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 9 | 5
Epigastric discomfort (Gastrointestinal disorders) | 0 | 2
Eructation (Gastrointestinal disorders) | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 1 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 11 | 7
Food poisoning (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 2
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 10 | 4
Gingival pain (Gastrointestinal disorders) | 2 | 1
Gingival recession (Gastrointestinal disorders) | 1 | 0
Gingival swelling (Gastrointestinal disorders) | 1 | 0
Gingivitis (Gastrointestinal disorders) | 3 | 0
Glossitis (Gastrointestinal disorders) | 2 | 1
Glossodynia (Gastrointestinal disorders) | 8 | 3
Haematochezia (Gastrointestinal disorders) | 3 | 5
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 5
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 3 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Oral discomfort (Gastrointestinal disorders) | 1 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 2 | 1
Perianal erythema (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 3 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 4 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 7 | 3
Rectal ulcer (Gastrointestinal disorders) | 1 | 0
Regurgitation (Gastrointestinal disorders) | 1 | 0
Salivary gland disorder (Gastrointestinal disorders) | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 2 | 0
Tooth discolouration (Gastrointestinal disorders) | 1 | 0
Tooth disorder (Gastrointestinal disorders) | 0 | 1
Tooth erosion (Gastrointestinal disorders) | 1 | 0
Tooth loss (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 3 | 12
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting projectile (Gastrointestinal disorders) | 0 | 1
Adverse drug reaction (General disorders) | 3 | 0
Application site irritation (General disorders) | 0 | 1
Atrophy (General disorders) | 0 | 1
Axillary pain (General disorders) | 2 | 1
Catheter site erythema (General disorders) | 1 | 1
Catheter site haematoma (General disorders) | 1 | 1
Catheter site inflammation (General disorders) | 1 | 1
Catheter site pain (General disorders) | 4 | 4
Catheter site rash (General disorders) | 0 | 1
Catheter site swelling (General disorders) | 0 | 1
Chest discomfort (General disorders) | 3 | 4
Cyst (General disorders) | 0 | 2
Device malfunction (General disorders) | 0 | 1
Device occlusion (General disorders) | 1 | 3
Disease progression (General disorders) | 0 | 3
Early satiety (General disorders) | 0 | 1
Extravasation (General disorders) | 1 | 0
Face oedema (General disorders) | 3 | 3
Feeling abnormal (General disorders) | 1 | 0
Feeling cold (General disorders) | 1 | 2
Feeling hot (General disorders) | 1 | 2
Fibrosis (General disorders) | 1 | 0
Gait disturbance (General disorders) | 3 | 8
Generalised oedema (General disorders) | 2 | 2
Gravitational oedema (General disorders) | 0 | 1
Hypothermia (General disorders) | 3 | 4
Ill-defined disorder (General disorders) | 2 | 1
Impaired healing (General disorders) | 2 | 1
Influenza like illness (General disorders) | 2 | 9
Infusion site extravasation (General disorders) | 0 | 1
Infusion site haematoma (General disorders) | 1 | 1
Infusion site pain (General disorders) | 1 | 0
Infusion site reaction (General disorders) | 1 | 0
Injection site haematoma (General disorders) | 0 | 1
Injection site reaction (General disorders) | 2 | 1
Irritability (General disorders) | 1 | 3
Local swelling (General disorders) | 2 | 0
Localised oedema (General disorders) | 1 | 1
Malaise (General disorders) | 3 | 5
Medical device complication (General disorders) | 0 | 1
Mucosal haemorrhage (General disorders) | 0 | 3
Mucosal hyperaemia (General disorders) | 0 | 1
Nodule (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 2
Temperature intolerance (General disorders) | 1 | 0
Tenderness (General disorders) | 0 | 1
Thirst (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Gallbladder fistula (Hepatobiliary disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 7 | 3
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1
Contrast media allergy (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 4 | 4
Hypersensitivity (Immune system disorders) | 7 | 7
Iodine allergy (Immune system disorders) | 0 | 1
Thrombosis in device (General disorders) | 5 | 3
Ulcer (General disorders) | 0 | 1
Multiple allergies (Immune system disorders) | 1 | 1
Seasonal allergy (Immune system disorders) | 6 | 6
Abscess (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Breast infection (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 7 | 5
Candidiasis (Infections and infestations) | 7 | 4
Catheter site cellulitis (Infections and infestations) | 0 | 1
Catheter site infection (Infections and infestations) | 4 | 6
Cellulitis (Infections and infestations) | 7 | 7
Cellulitis streptococcal (Infections and infestations) | 0 | 1
Chest wall abscess (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 2
Cystitis (Infections and infestations) | 5 | 5
Device related infection (Infections and infestations) | 4 | 5
Diverticulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 2 | 2
Escherichia sepsis (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 2 | 5
Folliculitis (Infections and infestations) | 4 | 8
Fungal infection (Infections and infestations) | 4 | 5
Fungal skin infection (Infections and infestations) | 2 | 2
Furuncle (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Genital herpes (Infections and infestations) | 1 | 0
Gingival infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 4
Hordeolum (Infections and infestations) | 1 | 2
Incision site infection (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 3 | 3
Influenza (Infections and infestations) | 4 | 3
Labyrinthitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 2 | 5
Localised infection (Infections and infestations) | 2 | 5
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 2 | 0
Mucocutaneous candidiasis (Infections and infestations) | 0 | 1
Nail bed infection (Infections and infestations) | 1 | 2
Nail bed infection bacterial (Infections and infestations) | 0 | 1
Nail infection (Infections and infestations) | 0 | 4
Nasopharyngitis (Infections and infestations) | 3 | 6
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 1 | 4
Oral candidiasis (Infections and infestations) | 2 | 1
Oral herpes (Infections and infestations) | 6 | 7
Oral infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 2 | 1
Parotitis (Infections and infestations) | 0 | 1
Pelvic abscess (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 4 | 2
Pneumonia (Infections and infestations) | 4 | 1
Rash pustular (Infections and infestations) | 2 | 3
Respiratory tract infection (Infections and infestations) | 0 | 3
Rhinitis (Infections and infestations) | 3 | 8
Sepsis (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 3 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 4 | 2
Tonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 5
Tooth infection (Infections and infestations) | 2 | 5
Viral infection (Infections and infestations) | 0 | 3
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 2 | 3
Vulvovaginitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 9 | 8
Excoriation (Injury, poisoning and procedural complications) | 2 | 2
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Eye penetration (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 7 | 6
Foot fracture (Injury, poisoning and procedural complications) | 1 | 2
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 2
Joint disclocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Open wound (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1
Vitreous injury (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 4
Wound complication (Injury, poisoning and procedural complications) | 3 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Bacterial test positive (Investigations) | 1 | 0
Blood albumin decreased (Investigations) | 2 | 1
Blood amylase increased (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 4 | 3
Blood chloride decreased (Investigations) | 1 | 1
Blood cholesterol increased (Investigations) | 1 | 1
Blood creatine increased (Investigations) | 0 | 1
Blood creatinine decreased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 10
Blood glucose decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 5 | 1
Blood homocysteine increased (Investigations) | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 0
Blood magnesium decreased (Investigations) | 3 | 4
Blood magnesium increased (Investigations) | 1 | 0
Blood parathyroid hormone increased (Investigations) | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 1
Blood phosphorus increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 3 | 1
Blood potassium increased (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 5
Blood sodium decreased (Investigations) | 2 | 1
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 1
Blood triglycerides increased (Investigations) | 0 | 2
Blood urea increased (Investigations) | 0 | 3
Blood uric acid increased (Investigations) | 0 | 2
Blood urine (Investigations) | 1 | 0
Body temperature increased (Investigations) | 1 | 0
Breath sounds abnormal (Investigations) | 5 | 1
Cardiac murmur (Investigations) | 0 | 2
Ejection fraction decreased (Investigations) | 5 | 8
Electrocardiogram QT prolonged (Investigations) | 0 | 2
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
Fungal test positive (Investigations) | 0 | 1
Gallop rhythm present (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Haematocrit decreased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 12 | 15
Haemoglobin increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 1
Heart rate irregular (Investigations) | 1 | 0
International normalised ratio (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 2 | 1
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 2 | 0
Neutrophil count (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 9 | 6
Neutrophil count increased (Investigations) | 0 | 2
Platelet count decreased (Investigations) | 7 | 2
Platelet count increased (Investigations) | 1 | 0
Protein total decreased (Investigations) | 0 | 1
Protein urine present (Investigations) | 1 | 0
Right ventricular systolic pressure increased (Investigations) | 0 | 1
Thyroxine increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 1
Urine leukocyte esterase positive (Investigations) | 0 | 1
Urine protein/creatinine ratio increased (Investigations) | 0 | 4
Vitamin D decreased (Investigations) | 1 | 2
Weight increased (Investigations) | 7 | 4
White blood cell count (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 7 | 9
White blood cell count increased (Investigations) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Enzyme abnormality (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1
Fluid intake reduced (Metabolism and nutrition disorders) | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 2 | 2
Folate deficiency (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 7 | 2
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 3
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 2 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 7
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 2 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ageusia (Nervous system disorders) | 1 | 1
Amnesia (Nervous system disorders) | 1 | 2
Aphasia (Nervous system disorders) | 3 | 1
Aphonia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 2 | 2
Balance disorder (Nervous system disorders) | 0 | 8
Burning sensation (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 0 | 1
Cranial nerve disorder (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Hyperaesthesia (Nervous system disorders) | 3 | 1
Hypersomnia (Nervous system disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 5 | 11
Hypogeusia (Nervous system disorders) | 1 | 2
Hyporeflexia (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 2
Memory impairment (Nervous system disorders) | 5 | 3
Migraine (Nervous system disorders) | 3 | 3
Nercolepsy (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Neurotoxicity (Nervous system disorders) | 5 | 4
Parosmia (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 2
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 2
Peroneal nerve palsy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0
Reflexes abnormal (Nervous system disorders) | 1 | 0
Restless legs syndrome (Nervous system disorders) | 3 | 6
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 2
Sensory disturbance (Nervous system disorders) | 0 | 1
Sinus headache (Nervous system disorders) | 6 | 8
Somnolence (Nervous system disorders) | 4 | 1
Speech disorder (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 3 | 2
Transient ischaemic attach (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 5 | 3
Visual field defect (Nervous system disorders) | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 1
Agitation (Psychiatric disorders) | 1 | 2
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 9 | 9
Depressed mood (Psychiatric disorders) | 2 | 1
Disorientation (Psychiatric disorders) | 2 | 1
Executive dysfunction (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 2 | 1
Mental status changes (Psychiatric disorders) | 6 | 1
Mood altered (Psychiatric disorders) | 2 | 7
Mood swings (Psychiatric disorders) | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 1
Nightmare (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 2
Stress (Psychiatric disorders) | 0 | 2
Bladder disorder (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 1
Chromaturia (Renal and urinary disorders) | 1 | 1
Cystitis interstitial (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 9 | 7
Haematuria (Renal and urinary disorders) | 1 | 7
Haemoglobinuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Incotinence (Renal and urinary disorders) | 0 | 2
Micturition urgency (Renal and urinary disorders) | 1 | 2
Nocturia (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 4
Proteinuria (Renal and urinary disorders) | 8 | 16
Renal failure (Renal and urinary disorders) | 1 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal pain (Renal and urinary disorders) | 1 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 4 | 4
Urinary retention (Renal and urinary disorders) | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Urogenital disorder (Renal and urinary disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 1
Breast induration (Reproductive system and breast disorders) | 1 | 0
Breast oedema (Reproductive system and breast disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 6 | 7
Breast tenderness (Reproductive system and breast disorders) | 1 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 2
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1
Genital lesion (Reproductive system and breast disorders) | 0 | 1
Genital rash (Reproductive system and breast disorders) | 0 | 1
Genital tract inflammation (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0
Oligomenorrhoea (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 2
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 2 | 1
Vaginal exfoliation (Reproductive system and breast disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 4 | 4
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0
Vaginal laceration (Reproductive system and breast disorders) | 2 | 0
Vaginal mucosal blistering (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 10
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 10
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 13
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Acne (Skin and subcutaneous tissue disorders) | 2 | 8
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 2 | 5
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 2
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 7 | 6
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 3 | 5
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 3
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hair colour changes (Skin and subcutaneous tissue disorders) | 2 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 6
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 2 | 3
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 | 0
Nail bed disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 10 | 7
Nail toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 6
Nipple ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 7
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 3
Onycholysis (Skin and subcutaneous tissue disorders) | 2 | 5
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 2
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Prurtitus generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
Purpura senile (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 3
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 4
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 1
Scab (Skin and subcutaneous tissue disorders) | 1 | 1
Scar (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 7 | 7
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 7 | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 7
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 5 | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Skin tightness (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 3
Swelling face (Skin and subcutaneous tissue disorders) | 3 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 3
Yellow skin (Skin and subcutaneous tissue disorders) | 1 | 0
Mastectomy (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Atteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 6
Haematoma (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 2
Infarction (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 7 | 14
Orthostatic hypotension (Vascular disorders) | 2 | 1
Pallor (Vascular disorders) | 1 | 2
Peripheral coldness (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 2
Phlebitis superficial (Vascular disorders) | 0 | 1
Poor peripheral circulation (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Systolic hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2
Vasodilatation (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.